CLINICAL TRIAL: NCT06897670
Title: Identifying Cerebral Hemodynamic Patterns in Mood Disorders and Mild Cognitive Impairment: A Functional Near-Infrared Spectroscopy (fNIRS) Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Lapid, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 24-012395
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Mild Cognitive Impairment
Keywords: functional near-infrared spectroscopy; diagnostics; mood disorders; mild cognitive impairment
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Cognitive Dysfunction; Mood Disorders | interventions — Cerebrovascular Circulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Controls: o No past or current psychiatric or cognitive disorder.
  Interventions: Other: Observational assessment using functional near-infrared spectroscopy (fNIRS), a noninvasive, portable brain imaging tool that measures changes in brain blood flow and oxygen levels.
- Major Depressive Disorder: * Diagnosis of major depressive disorder, confirmed through clinical evaluation.
  * No history of bipolar disorder or psychotic symptoms.
  Interventions: Other: Observational assessment using functional near-infrared spectroscopy (fNIRS), a noninvasive, portable brain imaging tool that measures changes in brain blood flow and oxygen levels.
- Bipolar Disorder: o Diagnosis of bipolar disorder I or II, confirmed through clinical evaluation.
  Interventions: Other: Observational assessment using functional near-infrared spectroscopy (fNIRS), a noninvasive, portable brain imaging tool that measures changes in brain blood flow and oxygen levels.
- Mild Cognitive Impairment (MCI): * Pre-existing clinical diagnosis of mild cognitive impairment, supported by neuropsychological testing and/or MRI, PET scan data.
  * No history of major psychiatric disorders, such as major depression, bipolar disorder or schizophrenia.
  Interventions: Other: Observational assessment using functional near-infrared spectroscopy (fNIRS), a noninvasive, portable brain imaging tool that measures changes in brain blood flow and oxygen levels.

INTERVENTIONS:
Other: Observational assessment using functional near-infrared spectroscopy (fNIRS), a noninvasive, portable brain imaging tool that measures changes in brain blood flow and oxygen levels. — Functional near-infrared spectroscopy (fNIRS) transcutaneously measures changes in oxyhemoglobin in the prefrontal cortex using light detection. It is designed to measure variations in cerebral hemodynamics on a real-time basis by radiating a near light beam, at two wavelengths of 780nm and 850nm of laser, into the cerebral cortex.
  Participants will undergo a one-time functional near-infrared spectroscopy (fNIRS) procedure to measure cerebral hemodynamic patterns.
  * Resting-State Measurement: 5-10 min resting-state scans.
  * Task-Based Measurement: Participants will be shown an instruction video. Participants will complete a Verbal Fluency Task (VFT) during the fNIRS scan (15-20 min).
  * During the fNIRS scan, optional basic vital signs will be measured using respiratory belts, photoplethysmography (PPG), and electrocardiogram (ECG).
  * Each participant will complete 3 sets of resting-state and task-based measurements.
  Total estimated time for fNIRS assessment: 45-60 min.

SUMMARY:
The purpose of this research is to measure brain activity in individuals with mood disorders and memory problems using a simple, safe, and noninvasive method called functional near-infrared spectroscopy (fNIRS). By comparing brain activity across different groups and relating it to symptom severity, this study aims to improve our understanding of how these conditions affect the brain.

DETAILED DESCRIPTION:
This study will examine cerebral hemodynamic patterns in individuals with mood disorders (major depressive disorder and bipolar disorder) and cognitive disorders (mild cognitive impairment) using functional near-infrared spectroscopy (fNIRS). The primary goal is to compare hemodynamic patterns between these groups, while the secondary goal is to explore correlations between these patterns and symptom severity based on standardized clinical assessments. Additionally, electrophysiological data, including photoplethysmography (PPG) and electrocardiogram (ECG), will be analyzed to investigate autonomic nervous system activity and its relationship with cerebral hemodynamics.

ELIGIBILITY:
Inclusion Criteria

General Inclusion Criteria (across all diagnostic groups):

* 18 years and older
* Ability to provide written informed consent
* Adequate cognitive and language abilities to understand and complete study tasks, including clinical assessments and fNIRS procedures
* Confirmed clinical diagnosis of major depressive disorder, bipolar disorder, or mild cognitive impairment (MCI)
* Stable psychiatric or cognitive condition, without acute episodes requiring immediate intervention

Specific Inclusion Criteria (for diagnostic groups):

* Healthy control

  o No past or current psychiatric or cognitive disorder
* Major depressive disorder (MDD):

  * Diagnosis of major depressive disorder, confirmed through clinical evaluation.
  * No history of bipolar disorder or psychotic symptoms.
* Bipolar disorder:

  o Diagnosis of bipolar disorder I or II, confirmed through clinical evaluation.
* Mild Cognitive Impairment (MCI):

  * Pre-existing clinical diagnosis of mild cognitive impairment, supported by neuropsychological testing and/or MRI, PET scan data.
  * No history of major psychiatric disorders, such as major depression, bipolar disorder or schizophrenia.

Exclusion Criteria

General Exclusion Criteria (across all diagnostic groups):

* Active primary psychotic or substance use disorders (except nicotine dependence) within the past year
* Any severe or unstable medical condition that could interfere with participation or data collection
* Any active neurological condition (including seizure disorder, traumatic brain injury, stroke) that could affect cognitive functioning or brain imaging results
* Inability to comply with study procedures, including cognitive testing, fNIRS assessment, or other assessments required by the protocol
* Pregnant women will be excluded due to potential physiological changes that could affect study outcomes

Specific Exclusion Criteria (for diagnostic groups):

* Healthy control

  o Any past or current psychiatric or cognitive disorder
* Major depressive disorder (MDD):

  * Diagnosis of bipolar disorder or schizophrenia.
  * Brain stimulation therapy within the past 3 months.
* Bipolar disorder:

  o Diagnosis of schizophrenia or schizoaffective disorder.
* Mild Cognitive Impairment (MCI):

  * Diagnosis of dementia.
  * Significant cognitive impairment preventing understanding or completion of study tasks.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified from the Mayo Clinic outpatient clinics in the Departments of Psychiatry, Psychology, Neurology, and Primary Care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in oxyhemoglobin | Baseline, 60 minutes
  Changes in oxyhemoglobin will be measured with a functional near-infrared spectroscopy (fNIRS) device by radiating a near light beam, at two wavelengths of 780nm and 850nm of laser, into the cerebral cortex. Oxyhemoglobin results are reported as a percentage of oxygen-bound hemoglobin compared to the total hemoglobin in the blood.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) | Baseline
  A clinician-administered tool revaluating depression severity. The 17-item version assesses symptoms such as depressed mood, insomnia, and somatic complaints. Each item is scored on a 3- or 5-point scale, resulting in total scores that range from 0 to 52, with scores of 0-7 considered normal, 8-16 indicating mild depression, 17-23 moderate depression, and 24 or greater severe depression.
Young Mania Rating Scale (YMRS) | Baseline
  A clinician-rated scale administered to measure the severity of manic symptoms in participants diagnosed with bipolar disorder (during manic or hypomanic episodes). It includes 11 items assessing areas such as elevated mood, irritability, and hyperactivity. Each item is scored on a scale of 0 to 4 or 0 to 8, with total scores ranging from 0 to 60. Severity thresholds include no significant symptoms (≤12), mild mania (13-20), moderate mania (21-35), and severe mania (>35).
Clinical Global Impression-Bipolar (CGI-BP) | Baseline
  A clinician-rated measure that provides a global assessment of illness severity, improvement, and therapeutic response in individuals with bipolar disorder. It includes separate ratings for mania, depression, and overall illness on a 7-point scale, where 1 indicates "normal, not at all ill" and 7 indicates "among the most severely ill."
Mini-Mental State Examination (MMSE) | Baseline
  The Mini-Mental State Examination is used to assess domains such as orientation, attention, memory, language, and visuospatial skills. It has a maximum score of 30, with lower scores indicating greater cognitive impairment. Scores are typically categorized as no cognitive impairment (24-30), mild cognitive impairment (18-23), and severe cognitive impairment (0-17).
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The PHQ-9 is a self-report questionnaire used to measure the severity of depressive symptoms over the past two weeks. This questionnaire is used in our clinical practice and will be collected from patient only if not already completed. It consists of nine items, each scored on a scale from 0 ("Not at all") to 3 ("Nearly every day"), with total scores ranging from 0 to 27. Higher scores indicate greater symptom severity, categorized as minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe depression (20-27).
Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Neuropsychological Battery | Baseline
  The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) is a standardized cognitive assessment tool designed to evaluate cognitive decline, particularly in Alzheimer's disease (AD) and mild cognitive impairment (MCI). It includes measures of verbal fluency, word list learning, delayed recall, recognition memory, constructional praxis, and global cognition. The battery incorporates a 15-item abbreviation of the Boston Naming Task (J2) and a slightly modified version of the MMSE that does not use serial 7s (J3).

CONTACTS AND LOCATIONS:
Overall Officials: Maria I. Lapid, M.D., Principal Investigator — Mayo Clinic; Paul H. Min, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yucel MA, Selb JJ, Huppert TJ, Franceschini MA, Boas DA. Functional Near Infrared Spectroscopy: Enabling Routine Functional Brain Imaging. Curr Opin Biomed Eng. 2017 Dec;4:78-86. doi: 10.1016/j.cobme.2017.09.011. Epub 2017 Oct 6. PMID 29457144
- [Background] Piper SK, Krueger A, Koch SP, Mehnert J, Habermehl C, Steinbrink J, Obrig H, Schmitz CH. A wearable multi-channel fNIRS system for brain imaging in freely moving subjects. Neuroimage. 2014 Jan 15;85 Pt 1(0 1):64-71. doi: 10.1016/j.neuroimage.2013.06.062. Epub 2013 Jun 28. PMID 23810973
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Spearing MK, Post RM, Leverich GS, Brandt D, Nolen W. Modification of the Clinical Global Impressions (CGI) Scale for use in bipolar illness (BP): the CGI-BP. Psychiatry Res. 1997 Dec 5;73(3):159-71. doi: 10.1016/s0165-1781(97)00123-6. PMID 9481807
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064